CLINICAL TRIAL: NCT04513899
Title: Development of a Community-based HCV Treatment Completion Intervention Among HCV Positive Homeless Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, Los Angeles (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Adeline Nyamathi, Founding Dean and Distinguished Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-5832; R21MD013580 (NIH)
Record Dates: First submitted 2020-08-05; First posted 2020-08-14 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C Virus (HCV) Infection
MeSH Terms: conditions — Hepatitis C; Infections | interventions — Community Health Workers; Nurses; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker/Registered Nurse (CHW/RN) (Experimental): Nurse-led Community Health Worker (CHW/RN) program delivered DOT for HCV treatment.
  Interventions: Behavioral: Community health worker (CHW)/ registered nurse (RN) [CHW/RN]
- Clinic-based Standard of Care (cbSOC) (Active Comparator): Standard of care for HCV treatment delivered by a clinic-based MD or clinic-based NP at the clinic site
  Interventions: Behavioral: Clinic-based Standard of Care (cbSOC) Program (control group)

INTERVENTIONS:
Behavioral: Community health worker (CHW)/ registered nurse (RN) [CHW/RN] — A team of 2-3 CHWs and a research RN will deliver all components of the program including daily DOT delivery of Direct Acting Antiviral (DAA) and assess HCV side effects all under the guidance of their RN. Recruitment will be continuous: each CHW may be assigned up to 7-8 participants every 2-3 months until the target sample size (n=54 for the intervention group) is achieved. After the first dose of the DAA, the CHW will run a brief weekly 1:1 education and case management session over the 8 or 12 weeks (total 20 minutes). The CHW/RN team will assist the participant in picking up the monthly medication and storing the medication in a secure, locked cabinet at the research office. The CHW will rigorously track participants who have missed a dose, and will also be involved in facilitating medical, mental health, substance use, social service, legal appointments for participants, housing referrals, and accompany the participants to the appointments.
  Arms: Community Health Worker/Registered Nurse (CHW/RN)
Behavioral: Clinic-based Standard of Care (cbSOC) Program (control group) — This program will be delivered by a clinic-based MD or clinic-based NP at the clinic site. Evaluation Staff (ES) will be hired and trained to do the interviewing/survey administration and follow-ups at the clinic-based site. The clinic NP will conduct, per usual care at the study clinics, the education and monitoring of these participants who will interact with the clinic-based-MD and/or NP monthly over the 8 or 12-week program. Usual care will include: 1) HCV pre-treatment education; 2) two month supply of DAA; 3) monitoring adverse events; and 4) responding to questions on HCV. Referral to drug/alcohol and housing programs will be provided over the standard of care. The cbSOC participants will not receive the community delivery of the DAA, or case management, or accompaniment to needed services. The cbSOC Program will receive the medication on a monthly basis from the clinic MD or NP.
  Arms: Clinic-based Standard of Care (cbSOC)

SUMMARY:
This randomized controlled trial (RCT) will test the efficacy of a Community Health Worker/Registered Nurse (CHW-RN) HCV intervention for homeless individuals, many who are also drug users. The intervention will be designed during Phase I of the proposal using an iterative process between a Community Advisory Board (CAB) and focus groups. The CHW/RN intervention will occur over a 2 or 3 month (8-12 weeks) period depending on the Direct-Acting Antiviral (DAA) prescribed. Homeless adults assigned to the CHW/RN HCV treatment group will receive culturally-sensitive education, case management, and daily DOT delivery of DAA by an RN-guided CHW. The CHW will run a brief (20 min) weekly 1:1 education and 20 min case management session over the 8 or 12 weeks and will deliver all components of the program (which will be developed and refined during Phase I). The CHW-RN HCV intervention will be compared to a clinic-based standard of care group (cbSOC). Primary outcomes are the completion of the Direct-Acting Agent (DAA) treatment (month 2 or 3) and SVR12 Cure (month 5 or 6). Secondary outcomes are improved mental health status, decrease in substance use, and improved access to health care, and shelter stability at month 5 or 6.

DETAILED DESCRIPTION:
HCV infection disproportionately affects homeless and drug-using populations and represents a critical focus for effective HCV prevention at the individual and community level. Homeless persons have a 26 fold increase in HCV prevalence compared to the general population; particularly with injection drug use (IDU). In fact, 50-80% of HCV infection is among persons who inject drugs (PWID). Among homeless populations, risk factors for HCV include older age, IDU, needle sharing, previous incarceration, veteran status, fair-or-poor health status, and sharing toothbrushes. Among the 48% of HCV-infected homeless persons who did not inject drugs, correlates of HCV infection include older age, less education, use of drugs, and history of multiple tattoos. While HCV treatment for PWID can reduce HCV prevalence, despite recommended guidelines, only 1-6% of drug-using HCV-infected persons have received treatment. Among the homeless adults, factors associated with low HCV treatment completion include untreated mental illness, current substance use, unstable housing, and limited access to care. Although the new Direct Acting Agent (DAA) are costly, cure rates have risen to above 98%. Yet limited research has been conducted on DAA agents among drug-using homeless adults. Extending HCV treatment beyond the traditional tertiary care model and involving peer supports can facilitate access to HCV treatment. The scientific premise of this proposal is that homeless HCV positive adults often do not obtain/complete HCV treatment due to significant psychosocial barriers. Thus, developing and testing a strategy that combines treatment with psychosocial support would be expected to change this outcome. To our knowledge, no randomized controlled trial (RCT) has yet assessed the efficacy of a comprehensive community-based model that incorporates HCV and substance use treatment to address HCV among homeless persons, despite the critical need that exists. The proposed treatment concept - Community Health Worker/Registered Nurse (CHW-RN) - is innovative and helps HCV treatment reach beyond the clinic walls, directly into the community where the homeless reside, reducing barriers to treatment. Guided by our community-based model, the CHW/RN intervention will focus on improving social support, coping skills, problem-solving, self-management, physical and mental health, substance use, and stable housing.

The proposed study will contribute to our knowledge about culturally-sensitive strategies for HCV treatment among homeless adults, many of whom use drugs and alcohol. It will address a substantial health disparity in a historically underserved population, with broader implications for public health. While DAAs have not been assessed among homeless adults using RCTs, homeless persons who are active drug users, in particular, have had challenges with uptake and compliance of other HCV treatments. To our knowledge, no study has evaluated the effect of a CHW/RN HCV treatment program, delivered in the community where the participant lives, compared to a cbSOC model to assess HCV treatment completion and Sustained Virologic Response (SVR) after 12 weeks of treatment completion. For further innovation, we will now evaluate the extent to which the pathways posed by the CHSCP and similar models, including the BMVP affect health outcomes by adding to Aim 3 analyses an examination of mechanisms of therapeutic change by the mediating effects of improved psychosocial and structural factors (e.g. housing, social support, etc ) on improved rates of SVR12. Improved understanding of the mechanisms of effect will advance the understanding of these factors and their role in determining health outcomes. The proposed study will pretest an RN-guided, CHW-delivered, program wherein a CHW/RN program will be developed and pretested with the community through focus group methodology. The intervention will focus on improving the completion of HCV treatment, reducing drug and alcohol use, reducing mental illness, and improving housing stability. The findings of this study can lay the groundwork for a subsequent larger trial to test the efficacy of the developed CHW/RN program more broadly and may inform health policy that could encourage enrollment of this high-risk group into HCV treatment. Results may also inform future cost-effective, community-based interventions that could be scaled-up and disseminated more broadly. Employing a treatment-as-prevention focus of HCV transmission in the community is urgent since HCV among the homeless represents a reservoir for HCV infection in the general population.

ELIGIBILITY:
Inclusion Criteria:

* currently homeless. A homeless person is defined as anyone who spent the previous night in a public or private shelter, a place not meant for sleeping (van, car, public facility, abandoned building) or in outdoor areas.
* age 18 or older;
* willing and able to provide informed consent;
* able to complete the screener;
* willing to have blood tests to be screened for HCV and tested HCV antibody positive;
* APRI ≤ 0.7, no signs of advanced cirrhosis (jaundice, ascites, encephalopathy) and willing to undergo the abdominal US as the standard of care (at the clinic).
* history of substance use (past 5 years).

Exclusion Criteria:

* current ongoing treatment for HCV;
* current HBV infection;
* HIV infection and not receiving medications for HIV treatment;
* not speaking English or Spanish; and
* testing pregnant; and
* judged to be cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ADELINE M NYAMATHI, PhD, Principal Investigator — University of California, Irvine; Lillian Gelberg, MD, Principal Investigator — University of California, Los Angeles
Locations (7):
- United States (7):
  - Amity Foundation, Los Angeles, Los Angeles, California
  - Cardinal Manning Center, Los Angeles, Los Angeles, California
  - Downtown Women Center, Los Angeles, Los Angeles, California
  - Los Angeles Christian Health Centers (LACHC), Los Angeles, California
  - Union Rescue Mission, Los Angeles, California
  - Weingart Center, Los Angeles, Los Angeles, California
  - St. John's Well Child and Family Center (SJWCFC), PRIME Specialty Clinic, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nyamathi A, Salem BE, Lee D, Yu Z, Hudson A, Saab S, Shin SS, Jones-Patten A, Yadav K, Alikhani M, Clarke R, Chang A, White K, Gelberg L. Exploratory assessment: Nurse-led community health worker delivered HCV intervention for people experiencing homelessness. Public Health Nurs. 2023 Sep-Oct;40(5):641-654. doi: 10.1111/phn.13204. Epub 2023 May 2. PMID 37132164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Based on our protocol, after screening was conducted, all eligible participants (n = 10) were enrolled over the length of the study, and after informed consent was completed.
Groups:
- Experimental: Community Health Worker/Registered Nurse (CHW/RN): Nurse-led Community Health Worker (CHW/RN) program delivered DOT for HCV treatment.
  A team of 2-3 CHWs and a research RN delivered all components of the program including daily DOT delivery of Direct Acting Antiviral (DAA) and assessed HCV side effects, all under the guidance of their RN. Recruitment was continuous. After the first dose of the DAA, the CHW ran a brief weekly 1:1 education and case management session over the 8 or 12 weeks (total 20 minutes). The CHW/RN team stored the medication in a secure, locked cabinet at the research office. The CHW rigorously tracked participants who missed a dose, and were involved in facilitating medical, mental health, substance use, social service, legal appointments for participants, housing referrals, and accompany the participants to the appointments.
- Active Comparator: Clinic-based Standard of Care (cbSOC): Standard of care for HCV treatment delivered by a clinic-based MD or clinic-based NP at the clinic site
  This program was delivered by a clinic-based MD or clinic-based NP at the clinic site. Evaluation Staff (ES) were hired and trained to do the interviewing/survey administration and follow-ups at the clinic-based site. The clinic NP conducted, per usual care at the study clinics, the education and monitoring of these participants who interacted with the clinic-based-MD and/or NP monthly over the 8 or 12-week program. Usual care included: 1) HCV pre-treatment education; 2) two-three month supply of DAA; 3) monitoring adverse events; and 4) responding to questions on HCV. Referral to drug/alcohol and housing programs were provided over the standard of care. The cbSOC participants did not receive the community delivery of the DAA, or case management, or accompaniment to needed services. The cbSOC Program received the medication on a monthly basis from the clinic MD or NP.
Period: Overall Study
Arm/Group | Experimental: Community Health Worker/Registered Nurse (CHW/RN) | Active Comparator: Clinic-based Standard of Care (cbSOC)
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants randomized to a study arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC) | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (6.75) | 55.7 (10.1) | 53.3 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing HCV Treatment
Description: The number of participants completing HCV treatment (7 days per week x 2- or 3 month treatment of DAA) was measured by pill count to measure adherence in both groups. For the RN/CHW group, directly observed therapy was utilized where the CHW or RN delivered the medication daily and documented each time s/he observed the participant swallow a pill.
  For the cbSOC Program (control group), the clinic-based MD/NP conducted a pill count monthly, based on the medications left in the pill bottle each month the participant is scheduled to pick up the next supply
Time Frame: 2-3 months depending on which DAA drug was provided. Some required 2 months and others, 3 months.
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
Number analyzed (Participants) | 4 | 6
Participants | 3 | 6

2. Primary Outcome: Number of Participants Attaining SVR12 (Sustained Viral Response at 12 Weeks After Treatment Completion)
Description: The number of participants who attained SVR12 Cure (HCV RNA < 25 IU/ml, detectable or undetectable) as tested at 5 or 6-month follow-up (12 weeks after treatment completion)
Time Frame: 5 or 6 months
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
Number analyzed (Participants) | 4 | 6
Participants | 3 | 4

3. Secondary Outcome: Drug Use
Description: Assessed by drug items in the Texas Christian University (TCU) Screen V. Yes/No responses to substance dependency questions and the frequency of drug use based on a 5-point scale from 1 (never) to 5 (daily) was assessed for each drug used. The range of scores on the 11-item Yes/no questions analyzed ranged from ranges from 0 - 11; corresponding to the number of symptoms endorsed by the participant and the severity of SUD: Mild disorder (2-3 points), moderate disorder (4-5 points), or severe disorder (6 or more points). The total score was calculated by adding the scores for all questions and averaging for all the participants at each follow-up time point. Drug Use was assessed at "2 or 3" months and "5 or 6" months follow-up.
Time Frame: 2 or 3- and 5 or 6-month follow-up
Population: Complete case
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
Number analyzed (Participants) | 3 | 6
score on a scale
  2 or 3 month follow up | 5 (4) | 3.33 (3.88)
  5 or 6 month follow up: number analyzed (Participants) | 3 | 5
  5 or 6 month follow up | 2.7 (3.8) | 4.8 (5.0)

4. Secondary Outcome: Alcohol Use Disorders Identification Test-Concise (AUDIT-C)
Description: Assessed by a brief alcohol screening instrument The Alcohol Use Disorders Identification Test-Concise (AUDIT-C). AUDIT-C reliably identifies persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). The AUDIT-C has 3 questions and is scored on a scale of 0-12. Each AUDIT-C question has 5 answer choices valued from 0 points to 4 points. The higher the score the more severe is the alcohol disorder. The total score was calculated by adding the scores for all questions and averaging for all the participants at each follow-up time point Based on the duration of DAA prescribed for the HCV treatment, the follow-up period was at "2 or 3" months and "5 or 6" months.
Time Frame: Assessment at 2 or 3- and 5 or 6-month follow-up
Population: Complete case
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
Number analyzed (Participants) | 3 | 5
score on a scale
  2 or 3 month follow up: number analyzed (Participants) | 2 | 5
  2 or 3 month follow up | 1.5 (2.12) | 2.8 (3.03)
  5 or 6 month follow up | 0.33 (0.58) | 3.6 (4.8)

5. Secondary Outcome: CAGE Substance Abuse Screening Scale
Description: Assessed by CAGE an internationally used assessment instrument for identifying alcoholics. Item responses on the CAGE are scored 0 or 1. The total score was calculated by adding up the scores for all four questions and averaging for all the participants for each time point. A total score of 2 or greater is considered clinically significant and may indicate alcohol-related issues.
  Based on the duration of DAA prescribed for the HCV treatment, the follow-up period was at "2 or 3" months and "5 or 6" months.
Time Frame: 2 or 3- and 5 or 6-month follow-up
Population: Complete case
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
Number analyzed (Participants) | 3 | 5
score on a scale
  2 or 3 month follow up | 0.667 (1.15) | 0.4 (0.894)
  5 or 6 month follow up | 0 (0) | 0.8 (1.79)

6. Secondary Outcome: Depression
Description: Mental Health will be assessed by Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a self-administered depression module of the Patient Health Questionnaire (PHQ). It contains 9 questions that help identify patients with clinically meaningful symptoms of depression. Patient responses are scored 0-3 with 0 representing "not at all" and 3 indicating "nearly every day;" thus, the PHQ-9 contains a total score range of 0-27. The total score was calculated by adding the scores for all questions and averaging for all the participants at each follow-up time point. The higher the score, the more severe is the alcohol disorder.
  Based on the duration of DAA prescribed for the HCV treatment, the follow-up period was at "2 or 3" months and "5 or 6" months.
Time Frame: 2 or 3- and 5 or 6-month follow-up
Population: Complete case
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
Number analyzed (Participants) | 3 | 5
score on a scale
  2 or 3 month follow up | 8 (7.55) | 8 (3.39)
  5 or 6 month follow up: number analyzed (Participants) | 2 | 5
  5 or 6 month follow up | 2 (0) | 7.6 (7.5)

7. Secondary Outcome: Mental Health
Description: Mental Health was assessed by the Mental Health Inventory (MHI)-5; well-demonstrated reliability for detecting psychological disorders. The MHI-5 comprises five questions. There are six possible responses to the questions, scored between 1 and 6. The score for each individual therefore ranges between 5 and 30. This is then transformed into a variable ranging from 0-100 using a standard linear transformation. The higher the score, the better the perception of mental health.
  Based on the duration of DAA prescribed for the HCV treatment, the follow-up period was at "2 or 3" months and "5 or 6" months.
Time Frame: 2 or 3- and 5 or 6-month follow-up
Population: Complete case
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
Number analyzed (Participants) | 3 | 5
units on a scale
  2 or 3 month follow up | 65.3 (32.3) | 76 (18.8)
  5 or 6 month follow up | 45.3 (16.2) | 62.4 (17.8)

8. Secondary Outcome: Health Care Access
Description: Health Care Access will include number of participants who completed 2 or more visits for health care or social services during the 2-3 month and 5-6 month follow-up
Time Frame: 2 or 3- and 5 or 6-month follow-up
Population: Complete case
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
Number analyzed (Participants) | 3 | 5
Participants
  2-3 month follow-up | 3 | 0
  5-6 month follow-up | 3 | 1

9. Post Hoc Outcome: Shelter Stability
Description: Shelter Stability is defined by number of participants who reported living in a shelter or apartment at month 2 or 3 and 5 or 6 months follow-up. The number of participants at each time period and in each arm were totaled.
Time Frame: 2 or 3 months and 5 or 6 months
Population: Complete Case
Measure: Count of Participants; unit: Participants
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
Number analyzed (Participants) | 3 | 5
Participants
  2 or 3 months | 0 | 2
  5 or 6 months | 2 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Same definition as clinicaltrials.gov
Groups:
- Clinic-based Standard of Care (cbSOC): Standard of care for HCV treatment delivered by a clinic-based MD or clinic-based NP at the clinic site. "Other [Not Including Serious] Adverse Events were not monitored/assessed for cbSOC Arm"
  Clinic-based Standard of Care (cbSOC) Program (control group): This program will be delivered by a clinic-based MD or clinic-based NP at the clinic site. Evaluation Staff (ES) will be hired and trained to do the interviewing/survey administration and follow-ups at the clinic-based site. The clinic NP will conduct, per usual care at the study clinics, the education and monitoring of these participants who will interact with the clinic-based-MD and/or NP monthly over the 8 or 12-week program. Usual care will include: 1) HCV pre-treatment education; 2) two month supply of DAA; 3) monitoring adverse events; and 4) responding to questions on HCV. Referral to drug/alcohol and housing programs will be provided over the standard of care. The cbSOC participants will not receive the community delivery of the DAA, or case management, or accompaniment to needed services. The cbSOC Program will receive the medication on a monthly basis from the clinic MD or NP.
Arm/Group | Community Health Worker/Registered Nurse (CHW/RN) | Clinic-based Standard of Care (cbSOC)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 3/4 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Community Health Worker/Registered Nurse (CHW/RN) (N=4) | Clinic-based Standard of Care (cbSOC) (N=0)
Headache (Nervous system disorders) | 2 (13) | NA
Tiredness (General disorders) | 3 (11) | NA
Loss of appetite (General disorders) | 2 (8) | NA
Diarrhea (Gastrointestinal disorders) | 2 (2) | NA
Sleepiness (General disorders) | 1 (1) | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | NA
Lightheadedness (General disorders) | 2 (3) | NA
Bleeding or bruising more easily than normal (General disorders) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
A major limitation is the small sample size due in part to low enrollment of PEH testing presumptive positive in the study as well as low numbers of PEH testing HCV positive. Finally, another limitation is the lack of generalizability of the study to other settings, such as urban settings outside of Skid Row and rural area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT04513899/Prot_SAP_000.pdf